CLINICAL TRIAL: NCT02647385
Title: Pain Control in Breast Surgery: Analgesia, Opioid Consumption and Inflammatory Response Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Raquel Chacon Ruiz Martinez, MS, PhD, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSL 2015-90
Record Dates: First submitted 2015-12-28; First posted 2016-01-06 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Anesthesia
Keywords: serratus anterior plane block; pectoral nerve block; breast surgery; cancer; analgesia; inflammatory cytokines
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Agnosia | interventions — Dental Occlusion; Lidocaine; S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General Anesthesia (Experimental): Interventions: include pain assessment, inflammatory response and opioid consumption.
  Interventions: Drug: Block with lidocaine for SAM and PEC I block
- General Anesthesia SAM and PEC I block (Experimental): Interventions: include pain assessment, inflammatory response and opioid consumption.
  Interventions: Drug: Block with lidocaine for SAM and PEC I block

INTERVENTIONS:
Drug: Block with lidocaine for SAM and PEC I block — Patients could be submitted to general anesthesia or general anesthesia associated with SAM and PEC I block with lidocaine before mastectomy.
  Interventions: include pain assessment, inflammatory response and opioid consumption.
  Other Names: Neuropathic pain

SUMMARY:
The serratus anterior muscle plane (SAM) block associated with pectoral nerve block type I (PEC I) may be a safe and effective alternative for the intraoperative of breast surgery, since there is evidence of pain reduction. However, correlation between regional anesthesia, postoperative pain and inflammatory response in breast surgery has not been demonstrated. The aim of this study is to compare the standard intravenous analgesia versus systemic analgesia associated with the SAM block and PEC I during breath cancer surgery. The following parameters will be evaluated: consumption of opioid intra and post-operative; post-operative pain and release of plasma inflammatory cytokines. It is a clinical prospective, randomized and controlled study. 50 individuals will be randomly divided into two groups. A group of patients receive general anesthesia during surgery and intravenous analgesia after the surgery and another group will receive general anesthesia associated with SAM and PEC I block during intraoperative and postoperative systemic analgesia. The postoperative pain will be assessed using the Visual Analogue Scale pain in the recovery room and 24 hours after surgery. Blood sample will be collected for determination of serum cytokines before surgery and 24 hours after the surgery. Also, it will be evaluated the development of chronic neuropathic pain 12 months after mastectomy, the use of analgesic medication, quality of life, depressive symptoms, and the levels of interleukin (IL)-1 beta, IL-6, and IL-10 as predictors of pain and depression.

DETAILED DESCRIPTION:
In breast surgery, regional anesthesia associated with general anesthesia during surgery has shown great results for the post-operative pain management, prevention of tumor recurrence and development of neuropathic pain. It has been shown that regional anesthesia attenuates the inflammatory response and systemic changes postoperatively during breast surgeries. Thus, it is important to include an additional analgesic intervention in breast surgery in order to decrease the local inflammatory response and the postoperative pain. Thus, the serratus anterior muscle plane (SAM) block associated with pectoral nerve block type I (PEC I) may be a safe and effective alternative for the intraoperative of breast surgery, since there is evidence of pain reduction. However, correlation between regional anesthesia, postoperative pain and inflammatory response in breast surgery has not been demonstrated. The aim of this study is to compare the standard intravenous analgesia versus systemic analgesia associated with the SAM block and PEC I during breath cancer surgery. The following parameters will be evaluated: consumption of opioid intra and post-operative; post-operative pain and release of plasma inflammatory cytokines. It is a clinical prospective, randomized and controlled study. Also, it will be evaluated the development of chronic neuropathic pain 12 months after mastectomy, the use of analgesic medication, quality of life, depressive symptoms, and the levels of interleukin (IL)-1 beta, IL-6, and IL-10 as predictors of pain and depression. 50 individuals will be randomly divided into two groups. A group of patients receive general anesthesia during surgery and intravenous analgesia after the surgery and another group will receive general anesthesia associated with SAM and PEC I block during intraoperative and postoperative systemic analgesia. The postoperative pain will be assessed using the Visual Analogue Scale pain in the recovery room and 24 hours after surgery. Blood sample will be collected for determination of serum cytokines before surgery and 24 hours after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiology (ASA) Scale I and II patients
* Patients submitted to breast cancer
* informed consent signature

Exclusion Criteria:

* Patients with chronic pain
* Local anesthesia reaction/allergy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12; Primary Completion 2024-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Patient´s Pain assessment | 24 hours
  The postoperative pain will be assessed using the Visual Analogue Scale pain in the recovery room and 24 hours after surgery.

SECONDARY OUTCOMES:
Opioid consumption | 24 hours
  The opioid consumption will be evaluated during and 24h after breast surgery
Cytokines | 24 hours
  Blood sample will be collected for determination of serum cytokines before surgery and 24 hours after the surgery.
Development of chronic pain | 1 year
  The development of chronic pain 12 months after mastectomy will be evaluated using the following scales: Douleur Neuropathique-4 - DN-4 (scores 4 or more indicates neuropathic character), Numeric Rating Scale - NRS ranging from 0 (no pain) -10 (worst pain) and Short-Form Health Survey (SF-36) ranging from zero (worst) to 100 (best score).

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Fernando Reis, PhD, Study Director — Hospital Sirio-Libanes
Locations (1):
- Hospital Sírio-Libanês, São Paulo, Brazil

REFERENCES:
- [Background] Buckley A, McQuaid S, Johnson P, Buggy DJ. Effect of anaesthetic technique on the natural killer cell anti-tumour activity of serum from women undergoing breast cancer surgery: a pilot study. Br J Anaesth. 2014 Jul;113 Suppl 1:i56-62. doi: 10.1093/bja/aeu200. Epub 2014 Jul 9. PMID 25009196
- [Background] Munoz M, Rosso M, Casinello F, Covenas R. Paravertebral anesthesia: how substance P and the NK-1 receptor could be involved in regional block and breast cancer recurrence. Breast Cancer Res Treat. 2010 Jul;122(2):601-3. doi: 10.1007/s10549-010-0850-y. Epub 2010 Mar 24. No abstract available. PMID 20333544
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Result] Matsumoto M, Flores EM, Kimachi PP, Gouveia FV, Kuroki MA, Barros ACSD, Sampaio MMC, Andrade FEM, Valverde J, Abrantes EF, Simoes CM, Pagano RL, Martinez RCR. Benefits in radical mastectomy protocol: a randomized trial evaluating the use of regional anesthesia. Sci Rep. 2018 May 18;8(1):7815. doi: 10.1038/s41598-018-26273-z. PMID 29777144
- [Derived] Flores EM, Gouveia FV, Matsumoto M, Bonacif THFS, Kuroki MA, Antunes GF, Campos ACP, Kimachi PP, Campos DO, Simoes CM, Sampaio MMC, Andrade FEM, Valverde J, Barros ACSD, Pagano RL, Martinez RCR. One year follow-up on a randomized study investigating serratus anterior muscle and pectoral nerves type I block to reduced neuropathic pain descriptors after mastectomy. Sci Rep. 2023 Mar 21;13(1):4591. doi: 10.1038/s41598-023-31589-6. PMID 36944694